CLINICAL TRIAL: NCT01566825
Title: The Influence of Amitriptyline (Amitriptylin-CT 25 mg®) on Learning in a Visual Discrimination Task (Karni-Sagi-paradigm)
Brief Title: The Influence of Amitriptyline on Learning in a Visual Discrimination Task
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dieter Kunz, MD (Other)
Responsible Party: Sponsor-Investigator, Dieter Kunz, MD, Director of the Research Group Sleep Research and Clinical Chronobiology, Department of Physiology CBF, Charité - Universitätsmedizin Berlin, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple
Other Study IDs: AVDT
Record Dates: First submitted 2012-03-27; First posted 2012-03-29 (Estimated); Last update posted 2012-03-29 (Estimated); Status verified 2012-03

CONDITIONS: Healthy Subjects
Keywords: amitriptyline; sleep dependent memory consolidation
MeSH Terms: interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Amitriptyline (Active Comparator)
  Interventions: Drug: Amitriptyline
- white 8 mm Lichtenstein® (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Amitriptyline — amitriptyline 25 mg at 9:30 pm, day 10, and 50 mg at 1:30 am, day 11
  Other Names: Saroten
  Arms: Amitriptyline
Drug: Placebo — placebo(white 8 mm Lichtenstein®) at 9:30 pm, day 10, and at 1:30 am, day 11
  Arms: white 8 mm Lichtenstein®

SUMMARY:
The purpose of this study is to determine whether 75 mg amitriptyline affect the sleep dependent consolidation of procedural memory (visual discrimination task, Karni-Sagi-paradigm).

DETAILED DESCRIPTION:
Rapid eye movement (REM) sleep is considered critical to the consolidation of procedural memory - the memory of skills and habits. Many antidepressants strongly suppress REM sleep, however, and procedural memory consolidation has been shown to be impaired in depressed patients on antidepressant therapy. As a result, it is important to determine whether antidepressive therapy can lead to amnestic impairment. We thus investigate the effects of the anticholinergic antidepressant amitriptyline on sleep-dependent memory consolidation in 32 healthy men in a double-blind, placebo-controlled, randomized parallel-group study.

ELIGIBILITY:
Inclusion Criteria:

* male gender
* age 18 through 40 years
* ability to communicate effectively in German

Exclusion Criteria:

* shift work within the past 24 months
* any sleep disorder as measured by the Pittsburgh Sleep Quality Index
* irregular sleep/wake patterns or extreme chronotype as measured by the Morningness-Eveningness Questionnaire
* history of any neurologic or psychiatric disorders
* regular medication intake within the past four weeks
* contraindications for amitriptyline
* abnormal electrocardiogram (ECG)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2008-08; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
changes in the visual discrimination task's perception threshold | The visual discrimination task's perception treshold is assessed before sleep (day 10 at 6 pm) and after sleep (day 11 at 6 pm).
  Improvement in this task is defined as a decrease in the perception threshold between training and retrieval testing.

SECONDARY OUTCOMES:
amount of rapid eye movement (REM) sleep (sleep period time percentage) | night from day 10 to day 11

CONTACTS AND LOCATIONS:
Overall Officials: Dieter Kunz, MD, Study Chair — Charite University, Berlin, Germany; Dieter Kunz, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Charité - Universitätsmedizin Berlin, Department of Physiology CBF, Berlin, Germany

REFERENCES:
- [Derived] Goerke M, Cohrs S, Rodenbeck A, Kunz D. Differential effect of an anticholinergic antidepressant on sleep-dependent memory consolidation. Sleep. 2014 May 1;37(5):977-85. doi: 10.5665/sleep.3674. PMID 24790277